CLINICAL TRIAL: NCT00837252
Title: Pilot Study for the Evaluation of Finasteride in the Treatment of Chronic Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090075; 09-EI-0075 (Other: National Eye Institute IRB)
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Retinal Disease
Keywords: Central Serous Chorioretinopathy; Finasteride; Proscar; Retinal Eye Disease
MeSH Terms: conditions — Retinal Diseases; Central Serous Chorioretinopathy | interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Finasteride (Experimental)
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride — Participants received 5mg of oral finasteride daily for three months.
  Other Names: Propecia; Proscar

SUMMARY:
Central serous chorioretinopathy (CSC) is a retinal disorder characterized by an accumulation of serous fluid under the retina. Although acute CSC tends to spontaneously resolve on its own with minimal sequelae, chronic CSC tends to persist and lead to irreversible visual loss. The pathogenesis of CSC is complex; however, systemic androgens have been implicated. Finasteride is an anti-androgen medication that is widely used in the treatment of various conditions. The objective of this study was to investigate the safety and potential efficacy of oral finasteride as a treatment for chronic CSC.

Five participants with chronic CSC were enrolled into this uncontrolled, unmasked, Phase I/II study. An oral dose of finasteride, 5 mg daily, was administered to all participants for three months.

Following this, finasteride was withheld and participants were observed for another three months. If a participant experienced a beneficial effect during the period in which he received finasteride and then experienced a relapse during the observation period, finasteride was re-instituted for the remaining period of the study. Relapse was defined as a return to the baseline maximum lesion height and/or return to baseline lesion volume.

ELIGIBILITY:
Participant-Level Inclusion Criteria

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must be willing to undergo monthly pregnancy tests throughout the study.
4. Female participants of childbearing potential must agree to practice two* acceptable methods of birth control throughout the course of the study and for three months after their last oral dose of finasteride. Acceptable methods of birth control include hormonal contraception (birth control pills, injected hormones or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom and spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy in a partner).

   *Participants with hysterectomy or vasectomy are exempt from using two methods of birth control. However female participants with a tubal ligation are not exempt and are required to practice another acceptable method of birth control.
5. Participant agrees to take the appropriate precautions to ensure that persons who are pregnant, nursing or of childbearing potential do not handle the finasteride tablets.

Participant-Level Exclusion Criteria

1. Participant is in another investigational study and actively receiving study therapy.
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant has evidence of ocular disease other than CSC in either eye that may confound the outcome of the study (e.g., diabetic retinopathy with 10 or more hemorrhages or microaneurysms, uveitis, pseudovitelliform macular degeneration, moderate/severe myopia, etc.).
4. Participant has evidence of CNV.
5. Participant has abnormal liver function testing as defined by elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels that are greater than twice the respective upper limits of normal (ULN), i.e., ALT > 82 U/L and/or AST > 68 U/L. If a participant has ALT or AST levels greater than twice the ULN, the participant can be enrolled if cleared by hepatology.
6. Participant is expected to need ocular surgery during the course of the trial.
7. Participant is on steroid medication (oral, topical or inhaled).
8. Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve.
9. Participant has a systemic condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

Study Eye Inclusion Criteria

1. Eligible participants must have chronic CSC in at least one eye as defined by all of the following criteria:

   1. The presence of subretinal fluid, as determined by spectral domain OCT, AND
   2. The subretinal fluid must have been present for at least three months, or there is a recurrence of subretinal fluid within the past three months, AND
   3. The presence of characteristic fluorescein angiographic or autofluorescence features of CSC, such as one or more pinpoint leaks and/or diffuse retinal pigment epitheliopathy. This eye will be referred to as the "study eye."
2. Participant must have a steady fixation in the study eye in the foveal or parafoveal area and media clear enough for good quality photographs.
3. Participant must have visual acuity between 20/25 and 20/400 in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine B Meyerle, MD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gomolin JE. Choroidal neovascularization and central serous chorioretinopathy. Can J Ophthalmol. 1989 Feb;24(1):20-3. PMID 2469527
- [Background] Tewari HK, Gadia R, Kumar D, Venkatesh P, Garg SP. Sympathetic-parasympathetic activity and reactivity in central serous chorioretinopathy: a case-control study. Invest Ophthalmol Vis Sci. 2006 Aug;47(8):3474-8. doi: 10.1167/iovs.05-1246. PMID 16877418
- [Background] Spahn C, Wiek J, Burger T, Hansen L. Psychosomatic aspects in patients with central serous chorioretinopathy. Br J Ophthalmol. 2003 Jun;87(6):704-8. doi: 10.1136/bjo.87.6.704. PMID 12770965
- [Result] Forooghian F, Meleth AD, Cukras C, Chew EY, Wong WT, Meyerle CB. Finasteride for chronic central serous chorioretinopathy. Retina. 2011 Apr;31(4):766-71. doi: 10.1097/IAE.0b013e3181f04a35. PMID 21273946

RESULTS

PARTICIPANT FLOW:
Groups:
- Finasteride: All five study participants (all of whom were diagnosed with chronic CSC) were administered a 5mg oral dose of finasteride daily for three months. After three months, the finasteride was withheld and the participants were observed for another three months.
Period: Overall Study
Arm/Group | Finasteride
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Finasteride
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Acuity at Month 3 Compared to Baseline.
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. This acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters the Snellen measurement is 20/20.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Finasteride
Number analyzed (Participants) | 5
ETDRS letters | 0 (22)

2. Secondary Outcome: Change in Visual Acuity at Month 6 Compared to Baseline
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Finasteride
Number analyzed (Participants) | 5
ETDRS letters | -3 (23)

3. Secondary Outcome: Change in Center-Subfield Macular Thickness at Month 3 Compared to Baseline
Description: Central-subfield macular thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Finasteride
Number analyzed (Participants) | 5
µm | -86 (105)

4. Secondary Outcome: Change in Center-Subfield Macular Thickness at Month 6 Compared to Baseline
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Finasteride
Number analyzed (Participants) | 5
µm | -69 (103)

5. Secondary Outcome: Change in Subretinal Fluid Volume at Month 3 Compared to Baseline
Description: Subretinal fluid volume was calculated after manually outlining the inner and outer borders of the subretinal fluid packet in the optical coherence tomography (OCT) images using the "Edit Segmentation" function of the Cirrus HD-OCT software. In cases where a pigment epithelial detachment was present, the volume of the pigment epithelial detachment was included in the calculation of subretinal fluid volume.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Finasteride
Number analyzed (Participants) | 5
µL | -0.58 (0.71)

6. Secondary Outcome: Change in Subretinal Fluid Volume at Month 6 Compared to Baseline
Description: as for outcome 5
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Finasteride
Number analyzed (Participants) | 5
µL | -0.53 (0.72)

7. Secondary Outcome: Change in Serum Dihydrotestosterone (DHT) Concentration at Month 3 Compared to Baseline
Description: The concentration of dihydrotestosterone (DHT) in blood serum was assessed from each participant at baseline and at Month 3. The mean change from baseline to Month 3 is reported here in picograms of DHT per milliliter of serum.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Finasteride
Number analyzed (Participants) | 5
pg/mL | -246 (116)

8. Secondary Outcome: Change in Serum Dihydrotestosterone (DHT) Concentration at Month 6 Compared to Baseline
Description: The concentration of dihydrotestosterone (DHT) in blood serum was assessed from each participant at baseline and at Month 6. The mean change from baseline to Month 6 is reported here in picograms of DHT per milliliter of serum.
Time Frame: 6 Months
Population: Only the 3 patients who were rechallenged with finasteride after Month 3 were included in this analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Finasteride
Number analyzed (Participants) | 3
pg/mL | -296 (87)

9. Secondary Outcome: Change in Serum Testosterone Level at Month 3 Compared to Baseline
Description: The concentration of testosterone in blood serum was assessed from each participant at baseline and at Month 3. The mean change from baseline to Month 3 is reported here in nanograms of testosterone per decaliter of serum.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Finasteride
Number analyzed (Participants) | 5
ng/dL | 0.38 (3.63)

10. Secondary Outcome: Change in Serum Testosterone Level at Month 6 Compared to Baseline
Description: The concentration of testosterone in blood serum was assessed from each participant at baseline and at Month 6. The mean change from baseline to Month 6 is reported here in nanograms of testosterone per decaliter of serum.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Finasteride
Number analyzed (Participants) | 5
ng/dL | -0.4 (3.38)

11. Secondary Outcome: Change in Urinary Cortisol Level at Month 3 Compared to Baseline
Description: The amount of cortisol found in urine was assessed from each participant at baseline and at Month 3. The mean change from baseline to Month 3 is reported here in micrograms.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Finasteride
Number analyzed (Participants) | 5
µg | 3 (24)

12. Secondary Outcome: Change in Urinary Cortisol Level at Month 6 Compared to Baseline
Description: The amount of cortisol found in urine was assessed from each participant at baseline and at Month 6. The mean change from baseline to Month 6 is reported here in micrograms.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Finasteride
Number analyzed (Participants) | 5
µg | -2 (18)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Finasteride
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finasteride (N=5)
Libido decreased (Psychiatric disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No